CLINICAL TRIAL: NCT01970384
Title: Transcranial Direct Current Stimulation for Dysphagia Therapy in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-140
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Stroke; Dysphagia
Keywords: transcranial direct current stimulation; stroke-related dysphagia; cortical plasticity
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial direct current stimulation (Experimental): 20 Minutes of transcranial direct current stimulation (20 min, 1 mA) administered over the contralesional cortical swallow motor area once daily over 4 consecutive days. In case of a brainstem stroke stimulation will be applied over the cortical swallow motor area of the right hemisphere.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): 20 Minutes of sham transcranial direct current stimulation (20 min, no current applied) administered over the contralesional cortical swallow motor area once daily over 4 consecutive days. In case of a brainstem stroke sham stimulation will be applied over the cortical swallow motor area of the right hemisphere.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — 20 Minutes of transcranial direct current stimulation (20 min, 1 mA) administered over the contralesional cortical swallow motor area once daily over 4 consecutive days. In case of a brainstem stroke stimulation will be applied over the cortical swallow motor area of the right hemisphere.
  Other Names: tDCS
  Arms: Transcranial direct current stimulation
Device: Sham stimulation — 20 Minutes of sham transcranial direct current stimulation (20 min, no current applied) administered over the contralesional cortical swallow motor area once daily over 4 consecutive days. In case of a brainstem stroke sham stimulation will be applied over the cortical swallow motor area of the right hemisphere.
  Other Names: sham tDCS
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to evaluate whether transcranial direct current stimulation of the cerebral swallow motor cortex in addition to standard care can enhance recovery of swallow function in acute dysphagic stroke patients compared to sham treatment plus standard care.

ELIGIBILITY:
Inclusion Criteria:

- dysphagia due to acute stroke

Exclusion Criteria:

* preexisting dysphagia
* comorbidities that can possibly cause dysphagia
* psychiatric comorbidities
* pacemaker or other implanted electronic devices
* inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
FEDSS (Fiberoptic Endoscopic Dysphagia Severity Scale) Score | Within three days after the last stimulation session

SECONDARY OUTCOMES:
Diet at discharge | by the time of discharge, an expected average of 2 weeks after the last stimulation session
Dysphagia Severity Rating Score | within three days after the last stimulation session
Endoscopically assessed swallow function | within three days after the last stimulation session
  Improvement of salient endoscopic findings

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Dziewas, PhD, Principal Investigator — Department of Neurology, University of Muenster
Locations (1):
- Department of Neurology, University of Muenster, Münster, Germany

REFERENCES:
- [Background] Suntrup S, Teismann I, Wollbrink A, Winkels M, Warnecke T, Floel A, Pantev C, Dziewas R. Magnetoencephalographic evidence for the modulation of cortical swallowing processing by transcranial direct current stimulation. Neuroimage. 2013 Dec;83:346-54. doi: 10.1016/j.neuroimage.2013.06.055. Epub 2013 Jun 23. PMID 23800793
- [Background] Dziewas R, Warnecke T, Olenberg S, Teismann I, Zimmermann J, Kramer C, Ritter M, Ringelstein EB, Schabitz WR. Towards a basic endoscopic assessment of swallowing in acute stroke - development and evaluation of a simple dysphagia score. Cerebrovasc Dis. 2008;26(1):41-7. doi: 10.1159/000135652. Epub 2008 May 30. PMID 18511871